CLINICAL TRIAL: NCT00598286
Title: Imaging of Cannabinoid CB1 Receptors Using [18F]FMPEP-d2
Brief Title: PET Imaging of Cannabinoid CB1 Receptors Using [18F]FMPEP-d2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Robert B. Innis, M.D./National Institute of Mental Health, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 080049; 08-M-0049
Record Dates: First submitted 2008-01-10; First posted 2008-01-21 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2012-05

CONDITIONS: CB1; Cannabinoid; PET; Brain Imaging
Keywords: CB1 Receptor; PET; Cannabinoid; [18F]FMPEP-d2; Brain Imaging; Healthy Volunteer; HV
MeSH Terms: interventions — 5-((3-fluoromethoxy)phenyl)-3-(1-phenylethylamino)-1-(4-trifluoromethylphenyl)pyrrolidin-2-one

INTERVENTIONS:
Drug: [18F]FMPEP-d2

SUMMARY:
The purpose of this protocol is to measure brain CB1 receptors in the hope to better understand how they work, so that one day we can understand how the CB1 receptors are involved in psychiatric, neurological, and behavioral disorders.

DETAILED DESCRIPTION:
BRAIN IMAGING

Objective

The central cannabinoid receptor (CB1) is one of the most abundant neuromodulatory receptors in the brain. It is found on glutamatergic, dopaminergic and GABA-ergic synaptic terminals and belongs to G-protein coupled receptor family. The CB1 is a target for drug therapy, including the use of an antagonist as an appetite suppressant. The central cannabinoid receptor CB1 has never been visualized in humans. In collaboration with Eli Lilly, we developed a promising PET ligand for the CB1 receptor: [18F]FMPEP-d2 ((3R,5R)-5-(3-(fluoromethoxy)phenyl)-3-((R)-1-phenylethylamino)-1-(4-(trifluoromethyl)phenyl)pyrrolidin-2-one).

Study Population

In the current protocol, we wish to evaluate [18F]FMPEP-d2 in approximately 10 healthy subjects.

Design

Brain imaging studies will consist of subject evaluation followed by PET and MRI scans.

Outcome Measures

We intend to determine the kinetics of brain uptake and washout, clearance in the plasma, and the distribution volume of [18F]FMPEP-d2 calculated with compartmental modeling. Distribution volume is proportional to the density of receptors and is equal to the ratio at equilibrium of uptake in brain to the concentration of parent radiotracer in plasma.

WHOLE BODY DOSIMETRY

Objective

Should the brain imaging studies prove to be successful, we will continue with whole body dosimetry studies. Preliminary dosimetry studies with [18F]d2-FMPEP have been performed in nonhuman primates; however, these need to be continued in humans before further investigation of this novel tracer can continue.

Study Population

In the current protocol, we wish to evaluate [18F]FMPEP-d2 in approximately 10 additional healthy subjects.

Design

The whole body dosimetry studies will consist of subject evaluation followed by a PET scan.

Outcome Measures

We intend to determine the whole body distribution of activity and thereby calculate radiation exposure to organs of the body.

BRAIN IMAGING WITH TEST/RE-TEST

Objective

Should the brain imaging and dosimetry studies prove to be successful, we will continue with test/retest brain imaging studies. Test/retest studies with [18F]FMPEP-d2 will provide evidence of reproducibility and strengthen the assurance that this radioligand can be used to assess pathology. Previous investigations in developing a CB1 receptor PET tracer have demonstrated the need to test reproducibility (Terry, In Writing; Burns et al 2007).

Study Population

In the current protocol, we wish to evaluate [18F]FMPEP-d2 in approximately 10 additional healthy subjects.

Design

The brain imaging test/retest studies will consist of subject evaluation followed by one MRI and two PET scans.

Outcome Measures

We intend to determine the reproducibility of the outcome measures from the brain imaging, namely, distribution volume.

ELIGIBILITY:
* INCLUSION CRITERIA:
* All subjects must be healthy and aged 18-65 years, with history/physical exam, ECG, and laboratory tests within one year of the PET scan.
* The volunteer must sign an informed consent form.

EXCLUSION CRITERIA:

* Current psychiatric illness, substance abuse including marijuana use, or severe systemic disease based on history and physical exam.
* Laboratory tests with clinically significant abnormalities or positive urine toxicology screen.
* Prior participation in other research protocols in the last year such that radiation exposure would exceed the annual limits.
* Pregnancy and breast feeding.
* Claustrophobia.
* Presence of ferromagnetic metal in the body or heart pacemaker.
* Positive HIV test.
* Employee of the investigative site or an immediate family member of an employee of the investigative site. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Employee of Eli Lilly and Company.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of novel PET tracer for CB1 in brain imaging.

SECONDARY OUTCOMES:
Distribution and variance of CB1 receptors in the brain of healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abi-Dargham A, Gandelman M, Zoghbi SS, Laruelle M, Baldwin RM, Randall P, Zea-Ponce Y, Charney DS, Hoffer PB, Innis RB. Reproducibility of SPECT measurement of benzodiazepine receptors in human brain with iodine-123-iomazenil. J Nucl Med. 1995 Feb;36(2):167-75. PMID 7830108
- [Background] Burger C, Buck A. Requirements and implementation of a flexible kinetic modeling tool. J Nucl Med. 1997 Nov;38(11):1818-23. PMID 9374364
- [Background] Burns HD, Van Laere K, Sanabria-Bohorquez S, Hamill TG, Bormans G, Eng WS, Gibson R, Ryan C, Connolly B, Patel S, Krause S, Vanko A, Van Hecken A, Dupont P, De Lepeleire I, Rothenberg P, Stoch SA, Cote J, Hagmann WK, Jewell JP, Lin LS, Liu P, Goulet MT, Gottesdiener K, Wagner JA, de Hoon J, Mortelmans L, Fong TM, Hargreaves RJ. [18F]MK-9470, a positron emission tomography (PET) tracer for in vivo human PET brain imaging of the cannabinoid-1 receptor. Proc Natl Acad Sci U S A. 2007 Jun 5;104(23):9800-5. doi: 10.1073/pnas.0703472104. Epub 2007 May 29. PMID 17535893
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2008-M-0049.html